CLINICAL TRIAL: NCT06726915
Title: Effect of Different Maternal Hemoglobin and Hematocrit Values on Perinatal Outcome
Status: Not yet recruiting | Type: Observational
Sponsor: Ali Mohamed Mohamed Ammar (Other)
Responsible Party: Sponsor-Investigator, Ali Mohamed Mohamed Ammar, Doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Anemia with pregnancy
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Hemoglobin and Hematocrit Values on Perinatal Outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the perinatal outcome in pregnancies with different levels of hemoglobin/hematocrit to verify which category of women should have iron supplementation if not all.

DETAILED DESCRIPTION:
Anaemia in pregnant women has been reported to have various adverse effects on both the mother and unborn foetus. These effects include preterm birth, a low birth weight and an increase in the risk of maternal and perinatal mortality . Postpartum anaemia impairs wound healing, increases the risk for readmission and/or prolonged hospitalization, and increases the cost of care for families .

Some investigators stated adverse perinatal outcome in pregnant mothers with high haemoglobin and haematocrit values and raised a question about the possible harmful effect of iron supplementation in such pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* 1. Pregnant women scheduled for labor or C.S (at term, 28-42 weeks). 3. Singleton pregnancy. 4. Age range: 18-40 years. 5. Willing to provide informed consent for participation and follow-up.

Exclusion Criteria:

1. Refusal to participate or consent.
2. Presence of non-iron deficiency anemia (e.g., hemoglobinopathies, chronic disease-related anemia).
3. Multiple pregnancies (e.g., twins or more).
4. Antepartum hemorrhage (e.g., placenta previa, placental abruption).
5. PAS.
6. Malformed fetus. -

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Pregnant female with age 18 to 40 year
Sampling Method: Non-Probability Sample
Enrollment: 403 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Fetal weight measurement- still birth or major morbidity | Baseline

SECONDARY OUTCOMES:
Maternal needs for iron therapy | Baseline
. Un-even postpartum period: Failure of lactation- DVT- CS wound complications Postpartum anaemia | Baseline

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Scholl TO. Iron status during pregnancy: setting the stage for mother and infant. Am J Clin Nutr. 2005 May;81(5):1218S-1222S. doi: 10.1093/ajcn/81.5.1218. PMID 15883455
- [Result] Blankson ML, Goldenberg RL, Cutter G, Cliver SP. The relationship between maternal hematocrit and pregnancy outcome: black-white differences. J Natl Med Assoc. 1993 Feb;85(2):130-4. PMID 8441188
- [Result] Lu ZM, Goldenberg RL, Cliver SP, Cutter G, Blankson M. The relationship between maternal hematocrit and pregnancy outcome. Obstet Gynecol. 1991 Feb;77(2):190-4. doi: 10.1097/00006250-199102000-00005. PMID 1988879
- [Result] Breymann C, Honegger C, Holzgreve W, Surbek D. Diagnosis and treatment of iron-deficiency anaemia during pregnancy and postpartum. Arch Gynecol Obstet. 2010 Nov;282(5):577-80. doi: 10.1007/s00404-010-1532-z. Epub 2010 Jun 25. PMID 20577752
- [Result] Pfeiffer CM, Looker AC. Laboratory methodologies for indicators of iron status: strengths, limitations, and analytical challenges. Am J Clin Nutr. 2017 Dec;106(Suppl 6):1606S-1614S. doi: 10.3945/ajcn.117.155887. Epub 2017 Oct 25. PMID 29070545